CLINICAL TRIAL: NCT00464568
Title: A Randomised, Open, Placebo-controlled 5-way Crossover Trial of Single Doses of Intranasal GSK256066 in Subjects With Seasonal Allergic Rhinitis (SAR).
Brief Title: A 5-way Treatment Period Trial of Single Doses of Intranasal GSK256066 in Patients With Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: IPR109764
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Results first posted 2017-08-21 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-07

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Seasonal allergic rhinitis,; hayfever
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — 6-((3-((dimethylamino)carbonyl)phenyl)sulfonyl)-8-methyl-4-((3-methyloxyphenyl)amino)-3-quinolinecarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK256066

SUMMARY:
This current study is planned as a dedicated pharmacodynamic (effect of drug on the body) study to investigate the dose response in rhinitic subjects at doses where GSK256066 has been proven to work (200mcg) or expected to (50mcg) work. This study also aims to investigate the lower end of the predicted therapeutic range.

ELIGIBILITY:
Inclusion Criteria:

* The subject is healthy.
* Body mass index less than 29.0 kg/m² , weight range of 55.0kg (females 50kg) to 95.0kg inclusive.
* They have a history of hayfever (repeated yearly episodes).
* They have a positive skin prick test for grass pollen at or within the 12 months preceding the screening visit.
* They have a positive radioallergosorbent test for grass pollen at or within the 12 months preceding the screening visit.
* non-smokers.
* They must have a baseline FEV1>80% predicted and a baseline FEV1(maximum recorded value)/ forced vital capacity (FVC) (maximum recorded value)>70%
* They are capable of giving informed consent
* They are available to complete all study measurements.

Exclusion Criteria:

* Pregnant or nursing females.
* Women of childbearing potential who are unwilling or unable to use an appropriate method of contraception.
* The subject has structural nasal abnormalities or nasal polyposis.
* Any respiratory disease other than mild stable asthma that is controlled with occasional use of as-needed short-acting beta-agonists and associated with normal lung function.
* The subject has a history of drug or other allergy that may contraindicate participation.
* The subject has participated in a study with a new molecular entity during the previous 4 months or in any clinical study in the previous 3 months
* The subject is concurrently participating in another clinical study and is exposed to an investigational or a non-investigational drug or device.
* The subject has a screening QTc value >450msec, PR interval outside the range 120 to 240msec or an ECG that is not suitable for QT measurements.In addition subjects will be excluded if they have a history of atrial and ventricular arrhythmia.
* The subject has a supine blood pressure that is persistently higher than 140/90 millimetres of mercury (mmHg) at screening.
* The subject has donated a unit of blood (450mL) within the previous 3 months or intends to donate within 3 months of completing the study.
* The subject is currently taking regular (or a course of) medication whether prescribed or not, including steroids, vitamins, and herbal remedies (e.g. St. John's Wort). Paracetamol (<2g/day) and occasional as needed use of short-acting beta agonists is permitted.
* Past or present disease which may affect study. outcome
* The subject regularly, or on average, drinks more than 4 units of alcohol per day - where 1 unit = ½ pint of beer (284mL), or 1 glass of wine (125mL), or 1 measure of spirit (25mL).
* The subject is at risk of non-compliance with the study procedures/restrictions.
* The subject has Hepatitis B, Hepatitis C, or HIV virus.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-03-28; Primary Completion 2007-05-16 (Actual); Study Completion 2007-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 32 healthy adult females and males aged 18 to 50 years and having a positive history of seasonal allergic rhinitis (SAR) were enrolled. The study was conducted at a single center in Germany from 28-March-2007 to 16-May-2007.
Pre-assignment Details: Participants who were positive for grass pollen on radioallergosorbent and skin prick testing were enrolled. Participants underwent Screening 7 to 28 days prior to study start.
Groups:
- Overall Study: Eligible participants received unit dose of nasal GSK256066 1 microgram (mcg) or 10 mcg or 50 mcg or 200 mcg or matching Placebo in any one of the five treatment periods in a randomized manner. Two treatment periods were separated by a 3 day washout period. Participants attended the unit on the morning of dosing and stayed until all study procedures were completed (approximately 4 hours) and were followed-up for maximum of 14 days.
Period: Overall Study
Arm/Group | Overall Study
Started | 32
Completed | 30
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Eligible participants received unit dose of nasal GSK256066 1 mcg or 10 mcg or 50 mcg or 200 mcg or matching Placebo in any one of the five treatment periods in a randomized manner. Two treatment periods were separated by a 3 day washout period. Participants attended the unit on the morning of dosing and stayed until all study procedures were completed (approximately 4 hours) and were followed-up for maximum of 14 days.
Arm/Group | Overall Study
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.7 (8.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 25
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White/Caucasian/European Heritage | 32

OUTCOME MEASURES:

1. Primary Outcome: Mean Messenger Ribonucleic Acid (mRNA) Concentrations as a Measure of Gene Expression
Description: The effect of GSK256066 on ribonucleic acid (RNA) levels indicative of Phosphodiesterase-4 (PDE4) inhibition in nasal scrape samples and on protein biomarkers of PDE4 inhibition in lavage samples was evaluated. Nasal lavage and scrapes were taken 2 to 3 hour post morning dose; bilateral nasal lavage was conducted before the scrape. Nasal scrape samples were taken from alternate nostrils. The novel RNA markers presented are cAMP responsive element modulator (CREM), dual specificity phosphatase 1(DUSP1), fos-like antigen 2(FOSL2), insulin receptor substrate 2 (IRS2), nuclear receptor subfamily 4, group A, member 2 (NR4A2), Phosphodiesterase-4A (PDE4A), Regulator of G-protein signalling 1 (RGS1), Serine/threonine protein kinase SNF1 like kinase (SNF1LK). Nasal lavage cytospins were stained with a SNF1LK specific monoclonal antibody by indirect immunofluorescence. Adjusted Geometric Mean and Standard error logs are presented.
Time Frame: Day 1
Population: All Subjects population comprised of all participants randomized to treatment who received at least one dose of study treatment (including placebo).
Measure: Geometric Mean (Standard Error); unit: COPIES/50 nanogram (NG)
Groups:
- Placebo: Eligible participants received a single dose of aqueous nasal spray of GSK256066 matching placebo via intranasal route, 1 puff per nostril and were followed-up up to maximum 14 days.
- GSK256066 1 mcg: Eligible participants received a single dose of GSK256066 1 mcg aqueous nasal spray via intranasal route, 1 puff of 0.5 mcg per nostril and were followed-up up to maximum 14 days.
- GSK256066 10 mcg: Eligible participants received a single dose of GSK256066 10 mcg aqueous nasal spray via intranasal route, 1 puff of 5 mcg per nostril and were followed-up up to maximum 14 days.
- GSK256066 50 mcg: Eligible participants received a single dose of GSK256066 50 mcg aqueous nasal spray via intranasal route, 1 puff of 25 mcg per nostril and were followed-up up to maximum 14 days.
- GSK256066 200 mcg: Eligible participants received a single dose of GSK256066 200 mcg aqueous nasal spray via intranasal route, 1 puff of 100 mcg per nostril and were followed-up up to maximum 14 days.
Arm/Group | Placebo | GSK256066 1 mcg | GSK256066 10 mcg | GSK256066 50 mcg | GSK256066 200 mcg
Number analyzed (Participants) | 31 | 30 | 32 | 30 | 31
COPIES/50 nanogram (NG)
  CREM | 2625.5 (0.03) | 2987.2 (0.03) | 3134.2 (0.03) | 3162.0 (0.03) | 3727.0 (0.03)
  DUSP1 | 8771.4 (0.04) | 12718.0 (0.04) | 13569.4 (0.04) | 15221.2 (0.04) | 15310.1 (0.04)
  FOSL2 | 10550.0 (0.03) | 15672.4 (0.03) | 16039.4 (0.03) | 17776.4 (0.03) | 16374.4 (0.03)
  IRS2 | 3260.5 (0.05) | 5052.0 (0.05) | 5059.6 (0.05) | 5671.2 (0.05) | 5083.8 (0.05)
  NR4A2 | 703.3 (0.07) | 1081.0 (0.07) | 1316.8 (0.07) | 1522.5 (0.07) | 1427.1 (0.07)
  PDE4A | 43.4 (0.05) | 44.5 (0.05) | 51.3 (0.05) | 51.7 (0.05) | 59.8 (0.05)
  RGS1 | 509.5 (0.06) | 542.2 (0.06) | 617.6 (0.06) | 698.4 (0.06) | 697.3 (0.06)
  SNF1LK | 2502.7 (0.05) | 6810.4 (0.05) | 7608.3 (0.05) | 8205.7 (0.05) | 8317.7 (0.05)
Statistical Analysis 1: Comparison: Placebo vs GSK256066 1 mcg; CREM; Placebo vs GSK256066 1 mcg; Test type: Superiority or Other; p = 0.1351, ANOVA; Treatment Ratios = 1.14, 95% CI 2-sided [0.96 to 1.35], Standard Error of Mean 0.037
Statistical Analysis 2: Comparison: Placebo vs GSK256066 10 mcg; CREM; Placebo vs GSK256066 10 mcg; Test type: Superiority or Other; p = 0.0383, ANOVA; Treatment Ratios = 1.19, 95% CI 2-sided [1.01 to 1.41], Standard Error of Mean 0.037
Statistical Analysis 3: Comparison: Placebo vs GSK256066 50 mcg; CREM; Placebo vs GSK256066 50 mcg; Test type: Superiority or Other; p = 0.0325, ANOVA; Treatment Ratios = 1.20, 95% CI 2-sided [1.02 to 1.43], Standard Error of Mean 0.037
Statistical Analysis 4: Comparison: Placebo vs GSK256066 200 mcg; CREM; Placebo vs GSK256066 200 mcg; Test type: Superiority or Other; p < 0.0001, ANOVA; Treatment Ratios = 1.42, 95% CI 2-sided [1.20 to 1.68], Standard Error of Mean 0.037
Statistical Analysis 5: Comparison: Placebo vs GSK256066 1 mcg; DUSP1; Placebo vs GSK256066 1 mcg; Test type: Superiority or Other; p = 0.0015, ANOVA; Treatment Ratios = 1.45, 95% CI 2-sided [1.16 to 1.82], Standard Error of Mean 0.049
Statistical Analysis 6: Comparison: Placebo vs GSK256066 10 mcg; DUSP1; Placebo vs GSK256066 10 mcg; Test type: Superiority or Other; p = 0.0002, ANOVA; Treatment Ratios = 1.55, 95% CI 2-sided [1.24 to 1.93], Standard Error of Mean 0.049
Statistical Analysis 7: Comparison: Placebo vs GSK256066 50 mcg; DUSP1; Placebo vs GSK256066 50 mcg; Test type: Superiority or Other; p < 0.0001, ANOVA; Treatment Ratios = 1.74, 95% CI 2-sided [1.38 to 2.17], Standard Error of Mean 0.050
Statistical Analysis 8: Comparison: Placebo vs GSK256066 200 mcg; DUSP1; Placebo vs GSK256066 200 mcg; Test type: Superiority or Other; p < 0.0001, ANOVA; Treatment Ratios = 1.75, 95% CI 2-sided [1.40 to 2.18], Standard Error of Mean 0.049
Statistical Analysis 9: Comparison: Placebo vs GSK256066 1 mcg; FOSL2; Placebo vs GSK256066 1 mcg; Test type: Superiority or Other; p = 0.0001, ANOVA; Treatment Ratios = 1.49, 95% CI 2-sided [1.22 to 1.81], Standard Error of Mean 0.043
Statistical Analysis 10: Comparison: Placebo vs GSK256066 10 mcg; FOSL2; Placebo vs GSK256066 10 mcg; Test type: Superiority or Other; p < 0.0001, ANOVA; Treatment Ratios = 1.52, 95% CI 2-sided [1.25 to 1.85], Standard Error of Mean 0.043
Statistical Analysis 11: Comparison: Placebo vs GSK256066 50 mcg; FOSL2; Placebo vs GSK256066 50 mcg; Test type: Superiority or Other; p < 0.0001, ANOVA; Treatment Ratios = 1.68, 95% CI 2-sided [1.38 to 2.05], Standard Error of Mean 0.043
Statistical Analysis 12: Comparison: Placebo vs GSK256066 200 mcg; FOSL2; Placebo vs GSK256066 200 mcg; Test type: Superiority or Other; p < 0.0001, ANOVA; Treatment Ratios = 1.55, 95% CI 2-sided [1.28 to 1.89], Standard Error of Mean 0.043
Statistical Analysis 13: Comparison: Placebo vs GSK256066 1 mcg; IRS2; Placebo vs GSK256066 1 mcg; Test type: Superiority or Other; p = 0.0034, ANOVA; Treatment Ratios = 1.55, 95% CI 2-sided [1.16 to 2.07], Standard Error of Mean 0.064
Statistical Analysis 14: Comparison: Placebo vs GSK256066 10 mcg; IRS2; Placebo vs GSK256066 10 mcg; Test type: Superiority or Other; p = 0.0029, ANOVA; Treatment Ratios = 1.55, 95% CI 2-sided [1.17 to 2.07], Standard Error of Mean 0.063
Statistical Analysis 15: Comparison: Placebo vs GSK256066 50 mcg; IRS2; Placebo vs GSK256066 50 mcg; Test type: Superiority or Other; p = 0.0003, ANOVA; Treatment Ratios = 1.74, 95% CI 2-sided [1.30 to 2.33], Standard Error of Mean 0.064
Statistical Analysis 16: Comparison: Placebo vs GSK256066 200 mcg; IRS2; Placebo vs GSK256066 200 mcg; Test type: Superiority or Other; p = 0.0027, ANOVA; Treatment Ratios = 1.56, 95% CI 2-sided [1.17 to 2.08], Standard Error of Mean 0.063
Statistical Analysis 17: Comparison: Placebo vs GSK256066 1 mcg; NR4A2; Placebo vs GSK256066 1 mcg; Test type: Superiority or Other; p = 0.0448, ANOVA; Treatment Ratios = 1.54, 95% CI 2-sided [1.01 to 2.34], Standard Error of Mean 0.092
Statistical Analysis 18: Comparison: Placebo vs GSK256066 10 mcg; NR4A2; Placebo vs GSK256066 10 mcg; Test type: Superiority or Other; p = 0.0033, ANOVA; Treatment Ratios = 1.87, 95% CI 2-sided [1.24 to 2.83], Standard Error of Mean 0.091
Statistical Analysis 19: Comparison: Placebo vs GSK256066 50 mcg; NR4A2; Placebo vs GSK256066 50 mcg; Test type: Superiority or Other; p = 0.0004, ANOVA; Treatment Ratios = 2.16, 95% CI 2-sided [1.42 to 3.30], Standard Error of Mean 0.092
Statistical Analysis 20: Comparison: Placebo vs GSK256066 200 mcg; NR4A2; Placebo vs GSK256066 200 mcg; Test type: Superiority or Other; p = 0.0010, ANOVA; Treatment Ratios = 2.03, 95% CI [1.34 to 3.08], Standard Error of Mean 0.091
Statistical Analysis 21: Comparison: Placebo vs GSK256066 1 mcg; PDE4A; Placebo vs GSK256066 1 mcg; Test type: Superiority or Other; p = 0.8718, ANOVA; Treatment Ratios = 1.03, 95% CI 2-sided [0.74 to 1.43], Standard Error of Mean 0.072
Statistical Analysis 22: Comparison: Placebo vs GSK256066 10 mcg; PDE4A; Placebo vs GSK256066 10 mcg; Test type: Superiority or Other; p = 0.3078, ANOVA; Treatment Ratios = 1.18, 95% CI 2-sided [0.86 to 1.63], Standard Error of Mean 0.071
Statistical Analysis 23: Comparison: Placebo vs GSK256066 50 mcg; PDE4A; Placebo vs GSK256066 50 mcg; Test type: Superiority or Other; p = 0.2909, ANOVA; Treatment Ratios = 1.19, 95% CI 2-sided [0.86 to 1.66], Standard Error of Mean 0.072
Statistical Analysis 24: Comparison: Placebo vs GSK256066 200 mcg; PDE4A; Placebo vs GSK256066 200 mcg; Test type: Superiority or Other; p = 0.0539, ANOVA; Treatment Ratios = 1.38, 95% CI 2-sided [0.99 to 1.91], Standard Error of Mean 0.071
Statistical Analysis 25: Comparison: Placebo vs GSK256066 1 mcg; RGS1; Placebo vs GSK256066 1 mcg; Test type: Superiority or Other; p = 0.7393, ANOVA; Treatment Ratios = 1.06, 95% CI 2-sided [0.74 to 1.54], Standard Error of Mean 0.081
Statistical Analysis 26: Comparison: Placebo vs GSK256066 10 mcg; RGS1; Placebo vs GSK256066 10 mcg; Test type: Superiority or Other; p = 0.2967, ANOVA; Treatment Ratios = 1.21, 95% CI 2-sided [0.84 to 1.74], Standard Error of Mean 0.080
Statistical Analysis 27: Comparison: Placebo vs GSK256066 50 mcg; RGS1; Placebo vs GSK256066 50 mcg; Test type: Superiority or Other; p = 0.0934, ANOVA; Treatment Ratios = 1.37, 95% CI 2-sided [0.95 to 1.98], Standard Error of Mean 0.081
Statistical Analysis 28: Comparison: Placebo vs GSK256066 200 mcg; RGS1; Placebo vs GSK256066 200 mcg; Test type: Superiority or Other; p = 0.0919, ANOVA; Treatment Ratios = 1.37, 95% CI 2-sided [0.95 to 1.97], Standard Error of Mean 0.080
Statistical Analysis 29: Comparison: Placebo vs GSK256066 1 mcg; SNF1LK; Placebo vs GSK256066 1 mcg; Test type: Superiority or Other; p < 0.0001, ANOVA; Treatment Ratios = 2.72, 95% CI 2-sided [2.11 to 3.51], Standard Error of Mean 0.056
Statistical Analysis 30: Comparison: Placebo vs GSK256066 10 mcg; SNF1LK; Placebo vs GSK256066 10 mcg; Test type: Superiority or Other; p < 0.0001, ANOVA; Treatment Ratios = 3.04, 95% CI 2-sided [2.37 to 3.90], Standard Error of Mean 0.055
Statistical Analysis 31: Comparison: Placebo vs GSK256066 50 mcg; RGS1; Placebo vs GSK256066 50 mcg; Test type: Superiority or Other; p < 0.0001, ANOVA; Treatment Ratios = 3.28, 95% CI 2-sided [2.54 to 4.23], Standard Error of Mean 0.056
Statistical Analysis 32: Comparison: Placebo vs GSK256066 200 mcg; RGS1; Placebo vs GSK256066 200 mcg; Test type: Superiority or Other; p < 0.0001, ANOVA; Treatment Ratios = 3.32, 95% CI 2-sided [2.59 to 4.27], Standard Error of Mean 0.055

2. Secondary Outcome: Mean Forced Expiratory Volume in One Second (FEV1)
Description: The FEV1 is the volume of air forcefully exhaled in 1 second. The highest FEV1 value amongst the three recorded FEV1 readings was used for all FEV1 calculations. FEV1 was recorded pre-dose and at follow-up.
Time Frame: Up to 9 weeks
Population: All subjects population.
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Placebo | GSK256066 1 mcg | GSK256066 10 mcg | GSK256066 50 mcg | GSK256066 200 mcg
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32
Liters (L) | 4.073 (0.9045) | 4.116 (0.8506) | 4.018 (0.8564) | 4.151 (0.8726) | 4.096 (0.8909)

3. Secondary Outcome: Mean Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP) Over Study Period
Description: Vital signs included SBP and DBP. SBP and DBP were measured pre-dose. The measurements were taken at 5 minutes interval during each treatment period. Vital signs measurements were made with the participant in a supine position having rested in this position for at least 5 minutes before the first reading at each time point. Measurements that deviated substantially from previous readings were repeated immediately.
Time Frame: Up to 9 weeks
Population: All subjects population.
Measure: Mean (Standard Deviation); unit: Millimetres of mercury (mmHg)
Arm/Group | Placebo | GSK256066 1 mcg | GSK256066 10 mcg | GSK256066 50 mcg | GSK256066 200 mcg
Number analyzed (Participants) | 31 | 30 | 32 | 30 | 31
Millimetres of mercury (mmHg)
  DBP | 70.8 (6.06) | 69.4 (6.33) | 69.2 (6.67) | 70.6 (7.24) | 68.9 (6.83)
  SBP | 117.0 (10.76) | 117.0 (10.34) | 113.8 (9.51) | 118.9 (10.91) | 115.1 (9.97)

4. Secondary Outcome: Mean Heart Rate Over Study Period
Description: Vital signs included heart rate. Heart rate was measured pre-dose. The measurements were taken at 5 minutes interval during each treatment period. Vital signs measurements were made with the participant in a supine position having rested in this position for at least 5 minutes before the first reading at each time point. Measurements that deviated substantially from previous readings were repeated immediately.
Time Frame: Up to 9 weeks
Population: All subjects population.
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Placebo | GSK256066 1 mcg | GSK256066 10 mcg | GSK256066 50 mcg | GSK256066 200 mcg
Number analyzed (Participants) | 31 | 30 | 32 | 30 | 31
Beats/minute | 58.8 (9.47) | 59.7 (9.10) | 57.9 (9.16) | 60.5 (12.34) | 57.8 (10.84)

5. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Values
Description: Electrocardiogram variables evaluated included PR interval, QRS duration, QT interval, QT corrected by Bazett's formula (QTcB), QT corrected by Fridericia's formula (QTcF) and RR interval. ECG was performed pre-dose, one hour and four hour post-dose. The ECG measurements were made with the participant in a supine position having rested in this position for at least 10 minutes before each time-point. Baseline was defined as the pre-dose measurement on Day 1. Change from Baseline was calculated by subtracting Baseline values from post-Baseline values
Time Frame: Baseline (Day 1) to 9 weeks
Population: All subjects population.
Measure: Mean (Standard Deviation); unit: Millisecond (msec)
Arm/Group | Placebo | GSK256066 1 mcg | GSK256066 10 mcg | GSK256066 50 mcg | GSK256066 200 mcg
Number analyzed (Participants) | 31 | 30 | 32 | 30 | 31
Millisecond (msec)
  PR Interval, 1 hour post-dose | -1.10 (6.650) | -0.87 (6.962) | -0.13 (9.157) | 1.73 (8.132) | 1.81 (8.553)
  PR Interval, 4 hour post-dose | -4.06 (7.857) | -5.87 (11.374) | -3.00 (7.379) | -2.40 (10.081) | -5.74 (9.560)
  QRS Duration, 1 hour post-dose | -0.77 (3.783) | -0.27 (2.449) | -0.50 (3.172) | -1.40 (2.931) | 0.06 (4.049)
  QRS Duration, 4 hour post-dose | -0.97 (3.996) | -0.93 (3.005) | -1.06 (3.835) | -1.40 (2.931) | 0.13 (4.440)
  QT Interval, 1 hour post-dose | 3.55 (10.865) | 11.67 (13.996) | 6.38 (13.645) | 8.93 (12.213) | 4.77 (11.851)
  QT Interval, 4 hour post-dose | -17.29 (16.113) | -11.40 (16.079) | -13.88 (12.638) | -15.07 (21.151) | -16.52 (18.147)
  QTcB, 1 hour post-dose | 0.58 (13.393) | 1.67 (11.689) | -2.94 (9.277) | 1.23 (14.555) | 1.03 (14.061)
  QTcB, 4 hour post-dose | -2.32 (14.063) | 0.30 (18.646) | -4.44 (13.361) | -1.27 (15.726) | -2.32 (12.621)
  QTcF, 1 hour post-dose | 1.41 (9.975) | 4.39 (8.874) | 0.40 (8.707) | 4.22 (10.710) | 2.37 (11.237)
  QTcF, 4 hour post-dose | -7.07 (11.240) | -3.99 (13.260) | -7.27 (10.288) | -5.42 (13.281) | -6.82 (10.284)
  RR Interval, 1 hour post-dose | 15.65 (93.021) | 58.51 (94.468) | 46.48 (72.070) | 30.62 (95.905) | 14.37 (100.749)
  RR Interval, 4 hour post-dose | -77.76 (104.801) | -52.34 (136.084) | -52.06 (90.711) | -73.88 (113.590) | -75.43 (101.077)

6. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant.
Time Frame: Up to 9 weeks
Population: All subjects population.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK256066 1 mcg | GSK256066 10 mcg | GSK256066 50 mcg | GSK256066 200 mcg
Number analyzed (Participants) | 31 | 30 | 32 | 30 | 31
Participants
  AE | 7 | 6 | 6 | 8 | 10
  SAE | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Hematology Values of Potential Clinical Concern
Description: Blood samples for hematology were taken before dosing. Whole blood samples were collected and processed according to the local procedures at site. The samples were transferred to the local laboratory for analysis. The participants with hematology of potential clinical concern are reported. The potential clinical concern ranges (low and high) were given as: for white blood cell count (clinical concern range: 3 to 20 giga cells/liter), neutrophils (normal range: 2.1 to 10.0 giga cells/liter), hemoglobin (clinical concern upper value: >180 grams/liter). Only those parameters for which at least one value of potential clinical concern was reported are summarized.
Time Frame: Up to 9 weeks
Population: All subjects population.
Measure: Number; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 32
Participants | 4

8. Secondary Outcome: Number of Participants With Clinical Chemistry Values of Potential Clinical Concern
Description: Blood samples for clinical chemistry were taken before dosing. Whole blood samples were collected and processed according to the local procedures at site. The samples were transferred to the local laboratory for analysis. The participants with clinical chemistry values of potential clinical concern are reported. The potential clinical concern ranges (low and high) were given as: for total bilirubin levels (clinical concern upper value: >31 micromole/liter) and inorganic phosphorus level (normal range: 0.7-1.5 millimole/liter).
Time Frame: Up to 9 weeks
Population: All subjects population.
Measure: Number; unit: Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 32
Participants | 4

9. Secondary Outcome: Area Under the Plasma Drug Concentration Versus Time Curve (AUC0-last) of GSK256066
Description: The pharmacokinetics (PK) of GSK256066 were assessed in plasma by determining AUC(0-last). All participants who received at least one dose of the active investigational product provided at least one sample for plasma PK analysis. Blood samples for PK were collected pre-dose, 15 minutes, 30 minutes, 1, 2, 3 and 4 hours post-dose and analyzed for GSK256066. AUC (0-last) was not calculable for any participant at 1 mcg GSK256066 dose.
Time Frame: Pre-dose, 15 minutes, 30 minutes, 1, 2, 3 and 4 hours post-dose on Day 1
Population: PK parameter population comprised of all participants from the PK Concentration population (comprised of all participants from the All Subjects population for whom blood or nasal samples were taken for assaying study drug) for whom PK parameters were available. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram*hour per milliliter (pg*hr/mL)
Arm/Group | GSK256066 1 mcg | GSK256066 10 mcg | GSK256066 50 mcg | GSK256066 200 mcg
Number analyzed (Participants) | 0 | 4 | 18 | 29
Picogram*hour per milliliter (pg*hr/mL) |  | 7.7 (58) | 14.7 (59) | 41.9 (97)

10. Secondary Outcome: AUC (0-last) of Active Metabolite GSK614917
Description: The PK of GSK256066 were assessed in plasma by determining AUC(0-last). All participants who received at least one dose of the study drug provided at least one sample for plasma PK analysis. AUC (0-last) was not calculable in any participant at the 1, 10 or 50 mcg GSK256066 dose.
Time Frame: Pre-dose, 15 minutes, 30 minutes, 1, 2, 3 and 4 hours post-dose on Day 1
Population: PK parameter population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg * hr/mL
Arm/Group | GSK256066 1 mcg | GSK256066 10 mcg | GSK256066 50 mcg | GSK256066 200 mcg
Number analyzed (Participants) | 0 | 0 | 0 | 18
pg * hr/mL |  |  |  | 12.7 (63.0)

11. Secondary Outcome: Maximum Observed Plasma Drug Concentration (Cmax) of GSK256066
Description: The PK of GSK256066 were assessed in plasma by determining Cmax. All participants who received at least one dose of the study drug provided at least one sample for plasma PK analysis. Blood samples for PK were collected pre-dose, 15 minutes, 30 minutes, 1, 2, 3 and 4 hours post-dose and analyzed for GSK256066.
Time Frame: Pre-dose, 15 minutes, 30 minutes, 1, 2, 3 and 4 hours post-dose on Day 1
Population: PK Parameter population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram per mililiter (pg/mL)
Arm/Group | GSK256066 1 mcg | GSK256066 10 mcg | GSK256066 50 mcg | GSK256066 200 mcg
Number analyzed (Participants) | 3 | 10 | 29 | 30
Picogram per mililiter (pg/mL) | 6.3 (198) | 5.1 (110) | 5.9 (70) | 20.4 (121)

12. Secondary Outcome: Cmax of Active Metabolite GSK614917
Description: The PK of GSK614917 were assessed in plasma by determining AUC(0-last). All participants who received at least one dose of the study drug provided at least one sample for plasma PK analysis. C max was not calculable for any participant at the 1 mcg GSK256066 dose.
Time Frame: Pre-dose, 15 minutes, 30 minutes, 1, 2, 3 and 4 hours post-dose on Day 1
Population: PK parameter population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | GSK256066 1 mcg | GSK256066 10 mcg | GSK256066 50 mcg | GSK256066 200 mcg
Number analyzed (Participants) | 0 | 3 | 6 | 24
pg/mL |  | 2.7 (47.6) | 2.4 (20.1) | 5.2 (62.4)

13. Secondary Outcome: Time to Maximum Observed Plasma Drug Concentration (Tmax) and Time to Last Observed Plasma Drug Concentration (Tlast) of GSK256066
Description: The PK of GSK256066 were assessed in plasma by determining Tmax and Tlast. All participants who received at least one dose of the study drug provided at least one sample for plasma PK analysis. Blood samples for PK were collected pre-dose, 15 minutes, 30 minutes, 1, 2, 3 and 4 hours post-dose and analyzed for GSK256066.
Time Frame: Pre -dose, 15 minutes, 30 minutes, 1, 2, 3 and 4 hours post-dose on Day 1
Population: PK Parameter population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | GSK256066 1 mcg | GSK256066 10 mcg | GSK256066 50 mcg | GSK256066 200 mcg
Number analyzed (Participants) | 3 | 10 | 29 | 30
Hour
  Tlast | 3.000 [0.25 to 3.98] | 2.000 [0.52 to 4.00] | 3.020 [2.00 to 4.37] | 4.000 [1.03 to 4.08]
  Tmax | 3.000 [0.25 to 3.98] | 2.000 [0.50 to 4.00] | 2.000 [1.00 to 3.03] | 2.000 [1.00 to 4.05]

14. Secondary Outcome: Tmax and Tlast of Active Metabolite GSK614917
Description: The PK of GSK614917 were assessed in plasma by determining Tmax and Tlast. All participants who received at least one dose of the study drug provided at least one sample for plasma PK analysis. Tmax and Tlast could not be determined for any participant at the 1 mcg GSK256066 dose.
Time Frame: Pre-dose, 15 minutes, 30 minutes, 1, 2, 3 and 4 hours post-dose on Day 1
Population: PK parameter population.
Measure: Median (Full Range); unit: Hour
Arm/Group | GSK256066 1 mcg | GSK256066 10 mcg | GSK256066 50 mcg | GSK256066 200 mcg
Number analyzed (Participants) | 0 | 3 | 6 | 24
Hour
  Tlast |  | 2.000 [0.52 to 3.98] | 2.510 [1.97 to 4.00] | 4.000 [2.98 to 4.08]
  Tmax |  | 2.000 [0.52 to 3.98] | 2.010 [1.97 to 4.00] | 3.000 [2.00 to 4.05]

15. Secondary Outcome: Nasal Lavage Concentrations of GSK256066
Description: Nasal lavage samples were taken 2 -3 hour post morning dose and analyzed for GSK256066. Quantifiable levels of GSK256066 were observed in nasal lavage samples obtained 2-3 hours post-dose.
Time Frame: Day 1
Population: PK concentration population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram/milliliter (pg/mL)
Arm/Group | Placebo | GSK256066 1 mcg | GSK256066 10 mcg | GSK256066 50 mcg | GSK256066 200 mcg
Number analyzed (Participants) | 31 | 30 | 32 | 30 | 31
Picogram/milliliter (pg/mL) | 6.460 (269.6) | 124.700 (165.1) | 457.370 (233.5) | 1046.088 (161.8) | 2226.638 (161.7)

16. Secondary Outcome: Mean Levels of Total Vasodilator Stimulated Phosphoprotein (VASP) Protein, Phosphorylated(Phospho)157 VASP (pVASP) and phospho239 VASP in Lavage Cells
Description: Nasal lavage were taken 2 to 3 hour post morning dose; bilateral nasal lavage was conducted before the scrape. Nasal lavage samples were analyzed to explore the effects of GSK256066 on novel protein biomarkers including pVASP. Markers indicative of PDE4 inhibition such as VASP protein levels and phospho157 VASP were also measured in this study, in lavage cells, following positive data in an enabling study which showed increases in such protein levels in participants with allergic rhinitis following a single intranasal dose of salbutamol. Nasal lavage data from earlier studies showed that pVASP157 is the best marker and not pVASP239. pVASP239 was therefore not collected or analyzed as planned.
Time Frame: Day 1
Population: All subjects population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | GSK256066 1 mcg | GSK256066 10 mcg | GSK256066 50 mcg | GSK256066 200 mcg
Number analyzed (Participants) | 31 | 30 | 32 | 30 | 31
Percentage
  VASP: number analyzed (Participants) | 31 | 30 | 32 | 29 | 31
  VASP | 3.5734 (7.5089) | 2.9960 (4.0191) | 3.0920 (4.4718) | 3.6985 (5.2735) | 2.2363 (3.3898)
  pVASP: number analyzed (Participants) | 30 | 27 | 31 | 27 | 30
  pVASP | 4.4913 (12.4942) | 1.8662 (3.6169) | 2.9963 (4.1263) | 2.6670 (4.9340) | 3.0254 (5.1593)
Statistical Analysis 1: Comparison: Placebo vs GSK256066 1 mcg; Placebo vs GSK256066 1 mcg: VASP; Test type: Superiority or Other; p = 0.647226, Mixed effects analysis of variance model; Mean treatment difference = -0.5545, Standard Deviation 7.79598
Statistical Analysis 2: Comparison: Placebo vs GSK256066 10 mcg; Placebo vs GSK256066 10 mcg: VASP; Test type: Superiority or Other; p = 0.95084, Mixed effects analysis of variance model; Mean treatment difference = -0.3816, Standard Deviation 9.00754 — The mean treatment difference was calculated as treatment minus placebo
Statistical Analysis 3: Comparison: Placebo vs GSK256066 50 mcg; Placebo Vs GSK256066 50 mcg: VASP; Test type: Superiority or Other; p = 0.53499, Mixed effects analysis of variance model; Mean treatment difference = 0.0256, Standard Deviation 9.24118 — The mean treatment difference was calculated as treatment minus placebo
Statistical Analysis 4: Comparison: Placebo vs GSK256066 200 mcg; Placebo vs GSK256066 200 mcg: VASP; Test type: Superiority or Other; p = 0.81527, Mixed effects analysis of variance model; Mean treatment difference = -1.3371, Standard Deviation 7.54590 — The mean treatment difference was calculated as treatment minus placebo
Statistical Analysis 5: Comparison: Placebo vs GSK256066 1 mcg; Placebo Vs GSK256066 1 mcg: pVASP; Test type: Superiority or Other; p = 0.32998, Mixed effects analysis of variance model; Mean treatment difference = -2.8053, Standard Deviation 10.88217 — The mean treatment difference was calculated as treatment minus placebo
Statistical Analysis 6: Comparison: Placebo vs GSK256066 10 mcg; Placebo vs GSK256066 10 mcg: pVASP; Test type: Superiority or Other; p = 0.65729, Mixed effects analysis of variance model; Mean treatment difference = -1.6602, Standard Deviation 12.30724 — The mean treatment difference was calculated as treatment minus placebo
Statistical Analysis 7: Comparison: Placebo vs GSK256066 50 mcg; Placebo vs GSK256066 50 mcg: pVASP; Test type: Superiority or Other; p = 0.89831, Mixed effects analysis of variance model; Mean treatment difference = 0.1560, Standard Deviation 4.73976 — The mean treatment difference was calculated as treatment minus placebo
Statistical Analysis 8: Comparison: Placebo vs GSK256066 200 mcg; Placebo vs GSK256066 200 mcg: pVASP; Test type: Superiority or Other; p = 0.84479, Mixed effects analysis of variance model; Mean treatment difference = -1.5165, Standard Deviation 12.70748 — The mean treatment difference was calculated as treatment minus placebo

ADVERSE EVENTS:
Time Frame: Up to 9 weeks
Description: On-treatment Serious adverse events (SAE) and non-serious adverse events (nSAE) are reported for the All Subjects population which comprised of all participants randomized to treatment who received at least one dose of study treatment (including placebo).
Groups:
- Placebo: Participants received a single dose of aqueous nasal spray of GSK256066 matching placebo via intranasal route, 1 puff per nostril. The total duration of the study per participant was approximately 8 to 9 weeks (up to 4 weeks Screening and 3 weeks dosing (including washout) plus a Follow-up visit at least 7 days (and no more than 14 days) after the last treatment.
- GSK256066 1 mcg: Participants received a single dose of GSK256066 1 mcg aqueous nasal spray via intranasal route, 1 puff of 0.5 mcg per nostril. The total duration of the study per participant was approximately 8 to 9 weeks (up to 4 weeks Screening and 3 weeks dosing (including washout) plus a Follow-up visit at least 7 days (and no more than 14 days) after the last treatment.
- GSK256066 10 mcg: Participants received a single dose of GSK256066 10 mcg aqueous nasal spray via intranasal route, 1 puff of 5 mcg per nostril. The total duration of the study per participant was approximately 8 to 9 weeks (up to 4 weeks Screening and 3 weeks dosing (including washout) plus a Follow-up visit at least 7 days (and no more than 14 days) after the last treatment.
- GSK256066 50 mcg: Participants received a single dose of GSK256066 50 mcg aqueous nasal spray via intranasal route, 1 puff of 25 mcg per nostril. The total duration of the study per participant was approximately 8 to 9 weeks (up to 4 weeks Screening and 3 weeks dosing (including washout) plus a Follow-up visit at least 7 days (and no more than 14 days) after the last treatment.
- GSK256066 200 mcg: Participants received a single dose of GSK256066 200 mcg aqueous nasal spray via intranasal route, 1 puff of 100 mcg per nostril. The total duration of the study per participant was approximately 8 to 9 weeks (up to 4 weeks Screening and 3 weeks dosing (including washout) plus a Follow-up visit at least 7 days (and no more than 14 days) after the last treatment.
Arm/Group | Placebo | GSK256066 1 mcg | GSK256066 10 mcg | GSK256066 50 mcg | GSK256066 200 mcg
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/32 | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 7/31 | 6/30 | 6/32 | 8/30 | 10/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=31) | GSK256066 1 mcg (N=30) | GSK256066 10 mcg (N=32) | GSK256066 50 mcg (N=30) | GSK256066 200 mcg (N=31)
Headache (Nervous system disorders) | 3 | 1 | 2 | 3 | 4
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Nasal necrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 2 | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Idioventricular rhythm (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Listless (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.